CLINICAL TRIAL: NCT04415645
Title: Phase 1, Open-Label Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of a Single Intravenous Dose of [14C]-VVZ-149 in Healthy Adult Male Subjects
Brief Title: Absorption, Metabolism, Excretion, and Mass Balance Study of [14C]-VVZ-149 in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VVZ149-HMB-P1-US101
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Healthy Adult Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VVZ-149 Injections (Experimental)
  Interventions: Drug: [14C]-VVZ-149

INTERVENTIONS:
Drug: [14C]-VVZ-149 — A single IV infusion of radio-labeled VVZ-149

SUMMARY:
This is an open-label, single-dose, absorption, metabolism, excretion, and mass balance study following a single IV infusion of [14C]-VVZ-149 in healthy adult male subjects. Whole blood, plasma, urine, and fecal samples will be analyzed for at least 72 hours following the start of infusion to measure total radioactivity and plasma drug concentrations.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy, adult, male, 19-55 years of age, inclusive
* Continuous non-smoker
* BMI ≥ 18.0 and ≤ 32.0 kg/m2
* Medically healthy with no clinically significant medical history or findings
* Must agree to adhere to the contraception requirements

Key Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease
* History or presence of alcohol or drug abuse within the past 2 years
* History, presence or evidence of cardiovascular, renal or hepatic impairment
* Less or abnormal bowel movements
* Unable to refrain from or anticipates the use of any prohibited drugs
* Recent donation of blood/plasma or significant blood loss
* Radiation exposure within 12 months
* Participation in another clinical study within 30 days

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Mass balance | Day 15
  Sum of the percent of the total radioactivity recovered in urine and feces relative to the administered radioactivity dose
Total radioactivity (TRA) concentration equivalents in plasma | Day 15
TRA concentration equivalents in urine | Day 15
TRA concentration equivalents in feces | Day 15
Drug concentrations in plasma | Hour 48

SECONDARY OUTCOMES:
Treatment-emergent adverse events | Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States